CLINICAL TRIAL: NCT07407374
Title: A Prospective Observational Cohort Study of Quality of Life, Body Image, and Sexual Function in Women With Postpartum Abdominal Wall Insufficiency Syndrome (PPAWIS) Using Patient-Reported Outcome Measures
Brief Title: Patient-Reported Outcomes in Women With Postpartum Abdominal Wall Insufficiency (PPAWIS)
Acronym: EMPOWER
Status: Not yet recruiting | Type: Observational
Sponsor: Swissmed Hospital (Other)
Collaborators: Medical University of Gdansk (Other); Śmietański Hernia Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: PPAWIS-01
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diastasis Recti and Weakness of the Linea Alba; Abdominal Wall Defect; Postpartum Complication; Abdominal Wall Anomaly
Keywords: PROMs; postpartum abdominal wall insufficiency; PPAWIS; patient-reported outcomes; sexual function; women's health; core stability; quality of life; abdominal wall reconstruction
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with PPAWIS (Routine Care): Participants are women diagnosed with postpartum abdominal wall insufficiency syndrome (PPAWIS) receiving routine clinical care as determined by the treating clinicians and patient preferences. Management include surgical approaches according to usual practice. No intervention is assigned by the research protocol. Patient-reported outcome measures are collected at baseline and during follow-up.
  Interventions: Other: Routine Clinical Care

INTERVENTIONS:
Other: Routine Clinical Care — No intervention is assigned by the research protocol. Clinical management is determined by clinicians and patients according to usual practice; the study collects patient-reported outcome measures longitudinally.

SUMMARY:
Postpartum abdominal wall insufficiency syndrome (PPAWIS) is a multidimensional condition that may affect physical function, quality of life, body image, and sexual health in women after childbirth. Anatomical findings alone do not fully explain symptom burden or patient experience.

This prospective observational cohort study will collect validated patient-reported outcome measures (PROMs) from women with PPAWIS receiving routine care. PROMs will be assessed at baseline and during follow-up to describe symptom burden and changes over time. The study aims to improve understanding of the patient-centered impact of PPAWIS and to support development of standardized assessment pathways in clinical practice.

DETAILED DESCRIPTION:
his is a prospective observational cohort study conducted in the setting of routine clinical care at Śmietański Hernia Center in Gdańsk (LUX MED Hospital) with collaboration from Medical University of Gdańsk. The study focuses on patient-centered outcomes in women with postpartum abdominal wall insufficiency syndrome (PPAWIS), a condition characterized by variable combinations of abdominal wall dysfunction and psychosocial impact after childbirth.

Participants will complete standardized, validated PROMs capturing quality of life, body image, and sexual function. Assessments will be performed at baseline (at/around qualification for routine care) and at predefined follow-up time points (e.g., 6 and 12 months). Clinical and demographic variables relevant for interpretation (e.g., time since last delivery, BMI, coexisting abdominal wall findings, and type of routine care received) will be recorded in a structured manner.

The study is non-interventional: treatment decisions and clinical management are determined by clinicians and patients according to usual practice and are not assigned by the research protocol. The primary purpose is to quantify baseline burden and describe longitudinal changes in PROMs, and to explore associations between patient-reported outcomes and selected clinical characteristics to inform future standardization of assessment and care pathways.

Data will be collected and stored using pseudonymized study identifiers. Participation is voluntary and can be withdrawn at any time without affecting clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-65 years
* Postpartum status: at least 6 months after last delivery
* Clinical diagnosis of postpartum abdominal wall insufficiency syndrome (PPAWIS), defined by abdominal wall dysfunction symptoms and/or significant quality-of-life impact, with supportive findings on physical examination and/or imaging (e.g., diastasis recti and/or related abdominal wall insufficiency features)
* Receiving routine clinical care for PPAWIS at the study site (surgical)
* Able and willing to provide informed consent and complete patient-reported outcome questionnaires at baseline and follow-up

Exclusion Criteria:

* Current pregnancy
* Planned pregnancy during the follow-up period (up to 12 months), if expected to interfere with outcome assessment
* Inability to complete questionnaires due to cognitive impairment or insufficient language proficiency in the validated questionnaire language version
* Severe uncontrolled psychiatric condition that, in the investigator's opinion, would prevent informed consent or reliable questionnaire completion
* Participation in another interventional study that could materially affect patient-reported outcomes related to abdominal wall function during the follow-up period

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18-65 years with postpartum abdominal wall insufficiency syndrome (PPAWIS), evaluated and managed in routine clinical care at the study site. Participants are assessed using validated patient-reported outcome measures at baseline and during follow-up to characterize symptom burden and changes over time.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life (WHOQOL-BREF) | Baseline and 6 months after baseline (window 5-7 months)
  Change from baseline in the WHOQOL-BREF domain scores and overall quality of life/health items in women with PPAWIS receiving routine care.

SECONDARY OUTCOMES:
Change in Sexual Function (FSFI) | Baseline and 6 months after baseline (window 5-7 months)
  Change from baseline in Female Sexual Function Index (FSFI) total score (and domains, if applicable).
Change in Body Image (Body Image scale) | Baseline and 6 months after baseline (window 5-7 months)
  Change from baseline in validated body image questionnaire score (instrument as specified in the study protocol and local language version).
Sustained Change in Quality of Life (WHOQOL-BREF) | Baseline and 12 months after baseline (window 11-13 months)
  Change from baseline in WHOQOL-BREF at long-term follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Śmietański, Prof., Principal Investigator — Śmietański Hernia Center, LUX MED Hospital in Gdańsk; Sylwia Jędrzejewska, MD, PhD, Study Chair — Polish Sexological Society

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in publications will be shared, including baseline and follow-up patient-reported outcome measure scores and a limited set of key clinical and demographic variables necessary to reproduce analyses (e.g., age range, BMI category, time since last delivery, presence of relevant abdominal wall findings). Direct identifiers will not be shared. Data will be pseudonymized and assessed for re-identification risk prior to release.
  Data will be shared for research purposes related to postpartum abdominal wall dysfunction and patient-reported outcomes, subject to approval of a qualified research proposal and execution of a data use agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD will be made available beginning 6 months after publication of the primary results and will remain available for 5 years.
Access Criteria: Access will be provided through controlled access. Requests must include a research proposal, analysis plan, and documentation of ethics approval (if applicable). Requests will be reviewed by the study steering group. Approved requestors will be required to sign a data use agreement specifying permitted uses, prohibiting re-identification attempts, and requiring secure data storage. Data will be shared in a de-identified format.

REFERENCES:
- [Background] Smietanski M, Smietanska IA, Zamkowski M. Post-partum abdominal wall insufficiency syndrome (PPAWIS): lessons learned from a single surgeon's experience based on 200 cases. BMC Surg. 2022 Aug 8;22(1):305. doi: 10.1186/s12893-022-01757-y. PMID 35941642